CLINICAL TRIAL: NCT06523023
Title: An Integrated Online Program Using Psychoeducation and Expressive Writing for People With Probable Post-traumatic Stress Disorder and Coexisting Dissociative Symptoms: a Pilot Randomised Controlled Trial
Brief Title: An Integrated Online Program Using Psychoeducation and Expressive Writing for People With Probable Post-traumatic Stress Disorder and Coexisting Dissociative Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Kam Ki Stanley, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21220891
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: post-traumatic stress; dissociation; structured writing; pilot study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Dissociative Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment will be ensured with the help of an independent statistician, who will be responsible for conducting the randomisation but will not be involved in any other parts of the project.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (an integrated online program) (Experimental): Our intervnetion is an integrated online program using psychoeducation and expressive writing. It is a 10-week program that consists of a 5-week psychoeducation module and a 5-week expressive writing module.
  Interventions: Behavioral: An integrated online program
- Waitlist control group (Other): After the treatment group has received and completed the integrated online program, the waitlist control group will receive the same program that is identical in content, procedures, and activities to the one received by the treatment group
  Interventions: Behavioral: An integrated online program

INTERVENTIONS:
Behavioral: An integrated online program — Our integrated online program combines validated psychoeducational materials on dissociation with components of strucutred writing therapy.

SUMMARY:
Objectives:

To evaluate the feasibility, acceptability, safety, and preliminary effects of an integrated online program with psychoeducation and expressive writing components for people with probable post-traumatic stress disorder (PTSD) and coexisting dissociative symptoms.

Hypotheses to be tested:

The program will be feasible, acceptable, and safe to participants. When compared with the waitlist control group, participants in the treatment group will report significantly lower PTSD symptom severity, lower dissociative symptom severity, and greater improvement on coping immediately post-intervention.

Design and subjects:

An assessor-blind, two-arm, randomised waitlist-controlled pilot study is proposed; 90 community adults with significant PTSD and dissociative symptoms will be recruited.

Instruments:

The PTSD Checklist 5, Dissociative Experiences Scale-Taxon, and Brief Coping Orientation to Problems Experienced inventory will be used. Semi-structured interviews will be conducted for process evaluation.

Intervention:

A 10-week integrated online program with psychoeducational and expressive writing components.

Main outcome measures:

The primary outcome is PTSD symptom severity. The secondary outcomes are dissociative symptom severity and coping. The feasibility, acceptability, and safety of the program will also be examined.

Data analysis: Feasibility and acceptability of the program will be assessed by examining the attrition rate, adherence rate, duration of subject recruitment, and post-program individual interviews. Generalised estimating equations with covariate adjustments will be used to examine the preliminary effects of the program.

Expected results:

Adults in the community who experienced significant PTSD and dissociative symptoms will become more resourceful to cope with their traumatic experiences and show more improvements on PTSD and dissociative symptoms.

ELIGIBILITY:
Inclusion Criteria:

(a) be Hong Kong Chinese residents between the ages of 18 and 65; (b) be able to read, write, and speak in Chinese/Cantonese; (c) meet the operational definitions of "probable PTSD" and "coexisting dissociative symptoms" in screening [score ≥31 on the Chinese version of the PTSD Checklist 5 (PCL-5) and ≥20 on the Chinese version of the Dissociative Experiences Scale-Taxon (DES-T)]; and (d) have access to a digital device with internet connectivity, such as a smartphone, tablet, or computer.

Exclusion Criteria:

(a) having participated in or currently receiving other psychoeducation/psychotherapies for PTSD or dissociative symptoms; (b) having clinically significant medical conditions that may interfere with safe study participation; (c) concurrent substance dependence, acute suicidality, psychosis, or gross cognitive impairment; and (d) visual, language, or communication difficulties.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder (PTSD) symptom severity | The outcome will be measured at baseline (T0) and immediately post-intervention (T1).
  The Chinese version PTSD Checklist 5 (PCL-5) will be used to measure DSM-5 PTSD symptom severity.

SECONDARY OUTCOMES:
Dissociative symptom severity | The outcome will be measured at baseline (T0) and immediately post-intervention (T1).
  The Chinese version Dissociative Experiences Scale-Taxon (DES-T) will be used to measure dissociative symptom severity.
Coping | The outcome will be measured at baseline (T0) and immediately post-intervention (T1).
  The Chinese version Brief Coping Orientation to Problems Experienced inventory (Brief-COPE) will be used to measure coping.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data generated and analysed during the current study will not be shared publicly. This decision is based on concerns regarding participant privacy and confidentiality, as well as the sensitive nature of the collected information. Therefore, the study's data will only be accessible to the research team and authorised personnel involved in the project.